CLINICAL TRIAL: NCT04252027
Title: Therapeutic Drug Monitoring of Fluconazole in Critically Ill Patients: a Longitudinal Follow-up of Trough Levels
Brief Title: Therapeutic Drug Monitoring of Fluconazole in Critically Ill Patients
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: S62242
Record Dates: First submitted 2020-01-28; First posted 2020-02-05 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Critically Ill Patients
Keywords: Pharmacokinetics; Fluconazole; Variability; Target attainment
MeSH Terms: interventions — Specimen Handling

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood and urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Sample collection — Plasma and urine sample collection

SUMMARY:
This prospective study will research the exposure and its variability to fluconazole after longitudinal administration in critically ill patients

DETAILED DESCRIPTION:
An open label, monocenter pharmacokinetic study will be carried out in critically ill patients, admitted at the University Hospitals Leuven, receiving multiple dose treatment with fluconazole.

The exposure to fluconazole in the ICU cohort over multiple days of treatment will be documented. Moreover, variability and the correlating covariates that can influence the fluconazole concentration, will be determined.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years
* Treatment with fluconazole
* Admitted to an ICU ward

Exclusion Criteria:

* < 18 years
* DNR 2 or 3

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill patients.
Sampling Method: Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2019-04-23 (Actual); Primary Completion 2020-03-05 (Actual); Study Completion 2020-03-05 (Actual)

PRIMARY OUTCOMES:
Exposure to fluconazole (trough levels) | On the day of sampling
  To document the trough levels (Cmin) of fluconazole in an ICU cohort over multiple days of treatment
Exposure to fluconazole (trough levels) | June 2020
  Determine if the Cmin target levels are attained.

SECONDARY OUTCOMES:
Variability in fluconazole trough levels | June 2020
  To determine the intra-and intersubject variability of the fluconazole trough levels
Influencing covariates | June 2020
  Determine possible covariates that might explain the fluconazole variability

CONTACTS AND LOCATIONS:
Overall Officials: Isabel Spriet, PharmD, PhD, Principal Investigator — UZ Leuven
Locations (1):
- UZ Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: Undecided